CLINICAL TRIAL: NCT06947824
Title: Effects of Fasted Morning vs. Evening Exercise on Post-Exercise Energy Intake
Brief Title: Time-of-Day Effects of Fasted Exercise on Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Karsten Koehler, Prof. Dr. Karsten Köhler, Technical University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MvE_FastEx
Record Dates: First submitted 2025-04-14; First posted 2025-04-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: Health; Energy Intake; Eating Behaviors; Appetite
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fasted Morning Exercise (12h AMEx) (Experimental): Exercise will take place in the morning, following a 12h overnight fast
  Interventions: Behavioral: Fasted Morning Exercise (12h)
- Fasted Evening Exercise (6h PMEx) (Active Comparator): Exercise will take place in the evening, following a 6h period of fasting
  Interventions: Behavioral: Fasted Evening Exercise (6h)
- Fasted Evening Exercise (12h PMEx) (Active Comparator): Exercise will take place in the evening, following a 12h period of fasting
  Interventions: Behavioral: Fasted Evening Exercise (12h)
- Fed Morning Exercise (AMEx Fed) (Active Comparator): Exercise will take place in the morning after consuming a small snack (30 min before exercise)
  Interventions: Behavioral: Fed Morning Exercise (AMEx Fed)
- Fed Evening Exercise (PMEx Fed) (Active Comparator): Exercise will take place in the evening after consuming a small snack (30 min before exercise)
  Interventions: Behavioral: Evening Fed Exercise (PMEx Fed)

INTERVENTIONS:
Behavioral: Fasted Morning Exercise (12h) — A 30-minute exercise session will take place on a treadmill in the morning (7:00, ~1h after participants' habitual wake-up time), after a 12h overnight fast. The session will consist of 30 minutes of steady state cycling at 65% of VO2max, following a 5 min warm-up.
  Arms: Fasted Morning Exercise (12h AMEx)
Behavioral: Fasted Evening Exercise (6h) — A 30-minute exercise session will take place on a treadmill in the evening (19:00, exactly 12 hours after the morning session), after a 6h fasting period. The session will consist of 30 minutes of steady state cycling at 65% of VO2max, following a 5 min warm-up.
  Arms: Fasted Evening Exercise (6h PMEx)
Behavioral: Fasted Evening Exercise (12h) — A 30-minute exercise session will take place on a treadmill in the evening (19:00, exactly 12 hours after the morning session), after a 12h fasting period. The session will consist of 30 minutes of steady state cycling at 65% of VO2max, following a 5 min warm-up.
  Arms: Fasted Evening Exercise (12h PMEx)
Behavioral: Fed Morning Exercise (AMEx Fed) — A 30-minute exercise session will take place on a treadmill in the morning (7:00, ~1h after participants' habitual wake-up time), after consuming a small pre-exercise snack (30 min before exercise). The session will consist of 30 minutes of steady state cycling at 65% of VO2max, following a 5 min warm-up.
  Arms: Fed Morning Exercise (AMEx Fed)
Behavioral: Evening Fed Exercise (PMEx Fed) — A 30-minute exercise session will take place on a treadmill in the evening (19:00, exactly 12 hours after the morning session), after consuming a small pre-exercise snack (30 min before exercise). The session will consist of 30 minutes of steady state cycling at 65% of VO2max, following a 5 min warm-up.
  Arms: Fed Evening Exercise (PMEx Fed)

SUMMARY:
This trial's aim is to investigate the time-of-day effects (morning vs. evening) of fasted exercise on acute and 24h post-exercise energy intake. Specifically, we will compare the effects of fasted morning exercise (12h overnight fast) vs. fasted (6h and 12h) evening exercise on total energy intake during a post-exercise ad libitum test meal as well as on 24h (free-living) energy intake. The secondary aim is to assess subjective appetite ratings before, immediately after, and 30 min post-exercise (visual analog scale). Healthy men and women aged 18-30 years will be included.

DETAILED DESCRIPTION:
In a five-way crossover design, participants will complete three fasted and one non-fasted exercise sessions on a treadmill in randomized order on weekdays with one week in between sessions: once in the morning (~1h after participants' habitual wake-up time) following a 12h overnight fast (12h AMEx), once in the evening (exactly 12h after the 12h AMEx condition) after a 6h fast (6h PMEx), and once in the evening (identical to the 6h PMEx condition) following a 12h fast (12h PMEx). As control conditions, a subsample of participants (n=17) will also complete a fed morning exercise condition (AMEx Fed; identical timing to 12h AMEx) and a fed evening exercise condition (PMEx Fed; identical timing to 12h PMEx), following a small pre-exercise snack (~10% of individual energy requirements; 30 min before exercise). The standardized meals provided before the fasting period contained 30% of the individual's daily energy requirements and consisted of ~50% carbohydrates, ~30% fat, and ~20% protein.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18.5.0-30.0 kg/m2
* weight stability (≤2.5 kg weight change during the past 3 months)
* ability to exercise at a vigorous intensity for 30 minutes

Exclusion Criteria:

* pregnancy or breastfeeding
* smoking
* history of or current eating disorders
* medical condition or use of medication that could affect appetite or pose any contraindications to exercise

As the menstrual cycle can cause fluctuations in food cravings and appetite, women of childbearing age were only eligible if they used hormonal contraceptives. To ensure constant exposure to exogenous estrogen and progestin throughout the study phase, participating women were further asked to use active hormone pills throughout the study period in both studies, a practice that is considered both safe and efficacious.

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Acute ad-libitum post-exercise energy intake (test meal) | 30 minutes after exercise
  Acute post-exercise energy intake (kcal) will be measured objectively using a single-item ad libitum test meal occurring 30 minutes after each exercise session. The meal will consist of cheese pizza, offered in excess of individual daily energy requirements, and all food will be provided at once.

SECONDARY OUTCOMES:
24h post-exercise energy intake | 24 hours post-exercise
  Post-exercise energy intake (ad libitum) will be self-reported (weighed food log) during the 24 hours following the exercise session. For the 6h PMEx and 12h PMEx conditions, this will encompass all food consumed after the exercise session until 19:00 the next day, including the test meal and typically the next day's breakfast, lunch, dinner, and all snacks consumed during this period. For the 12h AMEx condition, the 24-hour post-exercise period will encompass the test meal and typically lunch, dinner, snacks on the day of exercise, and the next day's breakfast, with the observation period ending at 07:00.
Subjective appetite measures | before exercise, immediately after exercise, and 30 minutes after exercise
  At each study condition visit, participants will rate their subjective perception of hunger, fullness, and desire to eat, and prospective food consumption on a 100mm visual analog scale anchored from "not at all" to "extremely" before each exercise session (Pre), immediately after (Post), and after an additional 30 minutes of post-exercise rest (Post30, immediately before the test meal),
Carbohydrate oxidation | continuously throughout the 30-minute exercise bout
  Carbohydrate oxidation, measured via indirect calorimetry
Fat oxidation | continuously throughout the 30-minute exercise bout
  Fat oxidation, measured via indirect calorimetry
Energy expenditure | continuously throughout the 30-minute exercise bout
  Energy expenditure, measured via indirect calorimetry

OTHER OUTCOMES:
Blood glucose | before exercise and immediately after exercise
  Blood glucose measured via capillary blodd (finger prick)
Blood lactate | before exercise and immediately after exercise
  measurement via capillary blood from the ear lobe
Breath ketones | before and immediately after exercise
  breath analysis via Lumen (MetaFlow Ltd) device
Blood ketones | before exercise and immediately after exercise
  measured via capillary blood (finger prick) and Freestyle Precision Neo (Abbott).

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request per the Technical University of Munich's data sharing policy.